CLINICAL TRIAL: NCT00479037
Title: A 24-week, International, Multi Centre, Randomised, Open Label, Parallel Group, Phase IV Clinical Trial Investigating Changes in Bone Formation Markers in Postmenopausal Women With Primary Osteoporosis Treated With Either PTH(1-84) or Strontium Ranelate
Brief Title: Effect of Full Length Parathyroid Hormone, PTH(1-84) or Strontium Ranelate on Bone Markers in Postmenopausal Women With Primary Osteoporosis (FP-006-IM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Nycomed
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FP-006-IM; 2006-006065-16
Record Dates: First submitted 2007-05-23; First posted 2007-05-25 (Estimated); Results first posted 2011-06-28 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Osteoporosis
Keywords: postmenopausal women with primary osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Parathyroid Hormone; strontium ranelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PTH(1-84) (Active Comparator)
  Interventions: Drug: Full Length Parathyroid Hormone, PTH(1-84)
- Strontium Ranelate (Active Comparator)
  Interventions: Drug: Strontium Ranelate

INTERVENTIONS:
Drug: Full Length Parathyroid Hormone, PTH(1-84) — Once daily subcutaneous injection in the abdomen by self administration
  Other Names: Preotact
  Arms: PTH(1-84)
Drug: Strontium Ranelate — The daily dose of 2 g (one sachet) strontium ranelate was to be mixed in a glass of water and taken immediately after mixing at bedtime at least 2 hours before or after intake of calcium, any food or drinks, other than water
  Arms: Strontium Ranelate

SUMMARY:
The primary objective of this trial is to show that PTH(1-84) is superior to strontium ranelate in bone formation measured as changes in bone formation markers over a treatment period of 24 weeks in postmenopausal women with primary osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women at or above the age of 50, diagnosed with primary osteoporosis may be enrolled in the trial if the following inclusion/exclusion criteria apply.

All inclusion criteria must be answered "yes" for a subject to be enrolled in the trial.

1. Has the subject given informed consent according to local requirements before any trial related activities? (A trial related activity is any procedure that would not have been performed during the routine management of the subject).
2. Is the subject female and at or above the age of 50?
3. Has the subject been postmenopausal for more than 5 years - in the judgement of the investigator?
4. Does the subject have primary osteoporosis and a T-score equal to or lower than -2.5 SD; T-scores must be assessed by DXA at the lumbar spine L1-L4, with a minimum of two assessable vertebrae, or at the total hip (right hip, if there is a right hip prosthesis, left hip can be used. If both hips are replaced the subject can be included with a lumbar scan only).
5. Is the subject currently taking calcium and vitamin D3 or is she willing to start such supplemental treatment and continue throughout the trial period, unless she develops hypercalcaemia?
6. Has the subject been taking supplemental calcium (1,000 mg) and vitamin D3 (800 IU) daily for at least 14 days (after screening) before blood sampling for eligibility evaluation? [*]
7. Is the subject able to self-inject PTH(1-84), or get the injections by a helper?

[*] Note that inclusion criteria no. 6 can not be evaluated at the time for screening, must be evaluated at randomisation, visit 2. See also exclusion criteria and note [**].

Exclusion criteria:

All exclusion criteria must be answered "no" for a subject to be enrolled in the trial.

Has the subject:

1. been treated with SERMS (selective oestrogen receptor modulators) or calcitonin within the last 1 month?
2. ever been treated with any bisphosphonate in intravenous form (i.v.)?
3. been treated with any bisphosphonates (alendronate, risedronate, or other bisphosphonates) for more than 3 years in total, or within the last 6 months?
4. been treated with fluoride for more than 3 months within the last 10 years?
5. ever been treated with strontium ranelate?
6. ever been treated with teriparatide or PTH(1-84)?
7. received or is the subject currently receiving chronic glucocorticosteroid treatment?

   Defined as more or equal to:

   5.0 mg prednisolon or equivalent daily for 3 months during the last year or 2.5 mg prednisolon or equivalent daily for 6 months during the last year. Local and inhalation steroids are permitted.
8. been treated for cancer (other than basocellular skin cancer) within the last 5 years?
9. ever received radiation therapy to the skeleton?
10. ever had malignant disease affecting the skeleton? or does the subject:
11. currently receive antiepileptic medication?
12. take any other medication (other than calcium and vitamin D3) that is known to affect bone metabolism? - according to the investigator's opinion.
13. have any known clinically significant diseases affecting calcium metabolism?
14. have any known history of metabolic bone diseases other than primary osteoporosis including hyperparathyroidism, Paget's disease, osteogenesis imperfecta, or osteomalacia)?
15. have any known history of hypersensitivity to parathyroid hormone or strontium or any of the excipients in the products?
16. have a serum vitamin D3, (serum 25(OH)D) level <20 ng/ml after at least 14 days of calcium and vitamin D3 supplementation? [**]
17. have a serum PTH of > 65 pg/ml and also a total serum calcium value >2.49 mmol/l? [**]
18. have hypercalcaemia (total serum calcium value >2.55 mmol/l), measured after at least 14 days of calcium and vitamin D3 supplementation? [**]
19. have elevated serum alkaline phosphatase? Defined as > 3X ULN [**]
20. have impaired kidney function with creatinine clearance < 30 ml/min (indirect measurement by serum creatinine)? [**]
21. have severe impaired liver function ? [**]
22. have phenylketonuria? or is the subject:
23. at risk of having venous thromboembolism including pulmonary embolism? - according to the investigator's opinion.
24. scheduled for vertebroplasty?
25. currently participating in a clinical trial with an investigational medical product, or has done so within the last 90 days, or plan to do so within the next 32 weeks? Previous and current participation in non-interventional trials is allowed.

[**] exclusion criteria no. 16 to 21 can not be evaluated before the result of the blood sampling (planned within the screening period and after at least 14 days of supplemental calcium/vitamin D3 intake) is available.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquarters
Locations (1):
- Nycomed, Roskilde, Denmark

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 82 subjects were randomized. Of these, one subject was randomized, but consent was withdrawn during the screening period; the subject did not receive any treatment. Therefore, the Intention to treat set (ITT) consisted of 81 subjects.
Groups:
- PTH(1-84): Once daily subcutaneous injection
- Strontium Ranelate: One sachet (2 g) per day, suspended in water
Period: Overall Study
Arm/Group | PTH(1-84) | Strontium Ranelate
Started | 41 | 40
Completed | 38 | 34
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTH(1-84) | Strontium Ranelate | Total
Number analyzed (Participants) | 41 | 40 | 81
Age Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.64) | 64.9 (8.49) | 64.4 (8.52)
Sex/Gender, Customized [Number; unit: participants]
  Female | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in the Bone Formation Marker N-terminal Propeptides of Human Procollagen Type I (P1NP) From Baseline to End of Trial
Description: P1NP is a bone formation marker that is derived from the amino-terminal propeptides of type I collagen and is considered a quantitative measure of newly formed type I collagen.
  Bone marker measurements were done by blood analysis.
Time Frame: Baseline and 24 weeks of treatment
Population: ITT (Intention to Treat) analysis. Number of participants analyzed = number of participants with data available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PTH(1-84) | Strontium Ranelate
Number analyzed (Participants) | 41 | 40
percent change | 446.1 (355.3) | -6.2 (36.9)
Statistical Analysis 1: Comparison: PTH(1-84) vs Strontium Ranelate; The bone marker values were log-transformed for the primary analysis as they were heavily skewed. Changes in log-transformed bone marker values were analyzed using an analysis of covariance (ANCOVA) with treatment and center as fixed effects and the baseline bone marker value as a covariate. An F-test was used to test the effect of treatment and the least square means were computed to assess the clinical difference between treatment groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values corresponding to the tests of treatment effect for the primary endpoints were adjusted using the Hochberg procedure; Mean Difference (Net) = 360.3, 95% CI 2-sided [256.5 to 494.3]

2. Primary Outcome: Percentage Change in the Bone Formation Marker Bone Specific Alkaline Phosphatase (BSAP) From Baseline to End of Trial
Description: BSAP is a marker of bone formation that reflects the cellular activity of osteoblasts.
  Bone marker measurements were done by blood analysis.
Time Frame: Baseline and 24 weeks of treatment
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PTH(1-84) | Strontium Ranelate
Number analyzed (Participants) | 41 | 40
percent change | 129.6 (100.3) | 4.9 (22.9)
Statistical Analysis 1: Comparison: PTH(1-84) vs Strontium Ranelate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 92.9, 95% CI 2-sided [63.8 to 127.1]

3. Secondary Outcome: Percentage Change in the Bone Resorption Marker C-Telopeptide Cross-links (CTX) From Baseline to End of Trial
Description: CTX is a marker of bone resorption, which is a degradation product of bone collagen.
  Bone marker measurements were done by blood analysis.
Time Frame: Baseline and 24 weeks of treatment
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PTH(1-84) | Strontium Ranelate
Number analyzed (Participants) | 41 | 40
percent change | 153.3 (132.4) | -3.7 (36.0)
Statistical Analysis 1: Comparison: PTH(1-84) vs Strontium Ranelate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value corresponding to the tests of treatment effect was adjusted using the Hochberg procedure; Mean Difference (Net) = 138.5, 95% CI 2-sided [94.8 to 191.8]

ADVERSE EVENTS:
Description: All safety analyses were based upon the safety set. The safety set consisted of all randomized subjects who had at least received one dose of trial drug
Arm/Group | PTH(1-84) | Strontium Ranelate
Serious Adverse Events (participants affected / at risk) | 2/40 | 2/40
Other Adverse Events (participants affected / at risk) | 29/40 | 19/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTH(1-84) (N=40) | Strontium Ranelate (N=40)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTH(1-84) (N=40) | Strontium Ranelate (N=40)
Nausea, mild severity (Gastrointestinal disorders) | 5 | 1
Nausea, moderate severity (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hypercalcaemia / mild severity (Metabolism and nutrition disorders) | 8 (9) | 0 (0)
Hypercalcaemia / moderate severity (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypervitaminosis D (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Headache, mild severity (Nervous system disorders) | 3 (3) | 2 (2)
Headache, moderate severity (Nervous system disorders) | 6 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 2 (2)
Malaise (General disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Venous insufficiency (Vascular disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
A limitation of the trial was the open label design, however this is not considered to affect the primary or secondary outcome of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After publication of the results or 24 months after Clinical Trial Report has been finalised, whichever comes first, Nycomed acknowledge the Investigator's rights to publish results from this trial. Any such scientific paper, presentation, communication, or other information concerning the investigation described in this protocol, must be submitted to Nycomed prior to submission for publication/presentation for review. Review comments will be given within a month from receipt of the manuscript.